CLINICAL TRIAL: NCT01357330
Title: A Phase 1 Dose Escalation Study of Combination Therapy With Oral SAR245408 (XL147) and Oral MSC1936369B in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Oral SAR245408 (XL147) and Oral MSC1936369B in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: TCD11742; U1111-1117-9893 (Other: UTN)
Record Dates: First submitted 2011-05-16; First posted 2011-05-20 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2012-08

CONDITIONS: Solid Tumors
Keywords: locally advanced or metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — XL147

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation (Experimental): Dose escalation phase The starting dose of SAR245408 will be 25-mg once daily (up to 200-mg). The starting dose of MSC1936369B will be 15- mg once daily (up to 90-mg)
  Interventions: Drug: SAR245408 (XL147); Drug: MSC1936369B

INTERVENTIONS:
Drug: SAR245408 (XL147) — Pharmaceutical form:capsule and tablet Route of administration: oral
Drug: MSC1936369B — Pharmaceutical form:capsule Route of administration: oral

SUMMARY:
Primary Objective:

- To determine the maximum tolerated dose(s) (MTD) and the recommended Phase 2 dose(s) (RP2D) of SAR245408 and MSC1936369B when combined in adult subjects with locally advanced or metastatic solid tumors.

Secondary Objective:

* To characterize the safety and tolerability of SAR245408 and MSC1936369B combination therapy administered orally to adult patients with locally advanced or metastatic solid tumors
* To evaluate the pharmacokinetic (PK) profile of SAR245408 and MSC1936369B when used in combination
* To evaluate the pharmacodynamic (PD) effect of the SAR245408/MSC1936369B combination by assessing target and pathway inhibition

DETAILED DESCRIPTION:
The duration of the study will include a period for screening of up to a maximum of 28 days, a pretreatment evaluation period of up to 5 days, the on-treatment period, followed by a minimum of 30-day follow-up after the last study drug administration.

The patient may continue study treatment until disease progression, unacceptable toxicity, or consent withdrawal.

The study will have 2 parts:

* Part one - Dose Escalation
* Part Two - Expansion. At the defined maximum tolerated doses (MTD(s), additional patients will be enrolled to collect safety, Pharmacokinetic, and Pharmacodynamic data

ELIGIBILITY:
Inclusion criteria:

Patient with advanced solid tumors for which there is no approved or curative therapy:

* has any advanced solid tumor with diagnosed alteration in 1 or more genes of the PI3K, and mitogen-activated protein kinase (MAPK) pathways and/or
* has a histologically or cytologically confirmed diagnosis of 1 of the following solid tumors: pancreatic, thyroid, colorectal, non-small cell lung, endometrial, renal, breast, ovarian carcinoma and melanoma

Exclusion criteria:

The patient has previously been treated with a PI3K inhibitor or a Mitogen-activated protein extracellular signal-regulated kinase (MEK) inhibitor

The patient has received:

* Chemotherapy, immunotherapy, hormonal therapy, biologic therapy, or any other anticancer therapy within 28 days or 5 half lives for noncytotoxics (whichever is shorter) of Day 1 of trial drug treatment (6 weeks for nitrosureas or mitomycin C)
* Any investigational agent within 28 days of Day 1 of trial drug treatment The patient is currently receiving anticoagulation therapy with therapeutic doses of warfarin (low-dose warfarin ≤1 mg/day, heparin, and low-molecular weight heparins are permitted) History of central nervous system metastases The patient has had congestive heart failure, unstable angina, a myocardial infarction, cardiac conduction abnormality or pacemaker or a stroke within 3 months of entering the study. The patient has retinal degenerative disease (hereditary retinal degeneration or age-related macular degeneration), history of uveitis, or history of retinal vein occlusion, or has medically relevant abnormalities identified on screening ophthalmologic examination.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Identification of maximum tolerated dose | up to 4 years

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events | up to 4 years
Pharmakokinetic parameters of SAR245408: Cmax | up to 4 years
Pharmakokinetic parameters of SAR245408: Tmax | up to 4 years
Pharmakokinetic parameters of SAR245408:AUCι | up to 4 years
Pharmakokinetic parameters of MSC1936369B: Cmax | up to 4 years
Pharmakokinetic parameters of MSC1936369B: Tmax | up to 4 years
Pharmakokinetic parameters of MSC1936369B: AUCι | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Investigational Site Number 840001, Boston, Massachusetts
  - Investigational Site Number 840002, Boston, Massachusetts
  - Investigational Site Number 840003, Nashville, Tennessee